CLINICAL TRIAL: NCT04899778
Title: Do Oral Contraceptives Protect Against Anterior Cruciate Ligament Injuries in Female Athletes
Brief Title: Do Oral Contraceptives Protect Against ACL Injuries in Female Athletes
Acronym: OC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Natasha Trentacosta, Surgeon, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00000922
Record Dates: First submitted 2021-05-17; First posted 2021-05-24 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Ligament Injury
Keywords: anterior cruciate ligament; birth control; oral contraceptive
MeSH Terms: interventions — Contraceptives, Oral; Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Contraceptive Pill (Experimental): Oral contraceptive, 1/day, for one year
  Interventions: Drug: Oral Contraceptive Pill, norethindrn a-e estradiol-iron
- No Oral Contraceptive (No Intervention): No intervention

INTERVENTIONS:
Drug: Oral Contraceptive Pill, norethindrn a-e estradiol-iron — tablet
  Other Names: Birth Control, norethindrn a-e estradiol-iron; Blisovi 24 Fe 1 mg-20 mcg
  Arms: Oral Contraceptive Pill

SUMMARY:
The purpose of this research study is to examine the impact of one type of commonly used birth control pill on blood levels of relaxin and measure changes in knee movement to determine whether there are changes in joint instability (indicating the knee is less stable) that may predispose female athletes to injury. Women not on hormonal birth control will also be enrolled to analyze differences between athletes on and not on birth control and to evaluate typical relaxin levels and knee laxity when birth control pills are not used.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Currently playing basketball, soccer, or volleyball at Loyola Marymount or Pepperdine
* If not currently on COC, regular menstrual cycle occurring every 21-35 days

Exclusion Criteria:

* Previous ACL injury
* Underlying neuromuscular disease
* Medical contraindication to COC use
* History of pregnancy
* Desire to conceive in the next year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Contraceptive Pill: Oral contraceptive, 1/day, for one year
  Oral Contraceptive Pill or IUC with hormones
Period: Overall Study
Arm/Group | Oral Contraceptive Pill | No Oral Contraceptive
Started | 31 | 42
Completed | 31 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- OCs Users: Participant athletes regularly took oral contraceptives or had a hormone-containing IUD.
- Non-OCs: Participant athletes were not on any form of contraception.
- Total: Total of all reporting groups
Arm/Group | OCs Users | Non-OCs | Total
Number analyzed (Participants) | 31 | 42 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 30 | 40 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (3.3) | 21.9 (3.7) | 21.6 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 42 | 73
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Injury
Description: Any injury resulting in time away from practice or competition
Time Frame: over the course of 1 year
Population: collegiate and professional female athletes
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Contraceptive Pill | No Oral Contraceptive
Number analyzed (Participants) | 31 | 42
Participants | 8 | 16

2. Secondary Outcome: Serum Relaxin Level
Description: level of relaxin measured in each subject
Time Frame: baseline, 4 month visit
Reporting Status: Not Posted, anticipated posting 2025-02

3. Secondary Outcome: Anterior Knee Laxity
Description: Anterior Knee laxity will be evaluated using the KT-2000 and measured in millimeters of anterior translation of the tibia relative to the femur
Time Frame: baseline, 4 month visit
Reporting Status: Not Posted

4. Secondary Outcome: Hip Rotation During a Single-legged Drop
Description: Hip flexion, adduction, and internal/external and coronal plane rotation of the knee measured during a singled-legged drop using motion tracking equipment.
Time Frame: baseline, 4 month visit
Reporting Status: Not Posted

5. Secondary Outcome: Knee Rotation During a Single-legged Drop
Description: as for outcome 4
Time Frame: baseline, 4 month visit
Reporting Status: Not Posted

6. Secondary Outcome: Joint Hypermobility
Description: Beighton score will be used to assess overall joint laxity. The Beighton score is on a nine-point scale that is based on 5 joint maneuvers. The maximum score is 9, which indicates increased laxity in the joints. A score of zero indicates inflexible joints.
Time Frame: baseline, 4 month visit
Reporting Status: Not Posted, anticipated posting 2025-04

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events were reported.
Groups:
- No Oral Contraceptive: No oral contraceptives used by athlete
Arm/Group | Oral Contraceptive Pill | No Oral Contraceptive
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/42
Other Adverse Events (participants affected / at risk) | 0/31 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT04899778/Prot_SAP_002.pdf